CLINICAL TRIAL: NCT04165564
Title: DECAMP 1 PLUS: Prediction of Lung Cancer Using Noninvasive Biomarkers
Status: Active, not recruiting | Type: Observational
Sponsor: Boston University (Other)
Collaborators: Johnson & Johnson (Industry); American College of Radiology Imaging Network (Network)
Responsible Party: Sponsor
Other Study IDs: H-39556
Record Dates: First submitted 2019-11-14; First posted 2019-11-18 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Pulmonary Disease
Keywords: Indeterminate pulmonary nodules; Molecular biomarkers for lung cancer diagnosis; Imaging for lung cancer diagnosis; High risk smokers
MeSH Terms: conditions — Lung Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Nasal brushing, Buccal scraping, Stool, Bronchial Biopsy, Bronchial brushing, Lung tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 - Screening: Participants in this group will be 55-77 years old and currently smoke or were former smokers with 30 pack-years or more (and quit less than 15 years ago)
  Interventions: Other: Institutional standard of care; Other: Biosamples of airway and blood
- Group 2 - Incidental: Participants in this group will be > 45 years old and currently smoke or were former smokers with 10 pack-years or more (and quit less than 15 years ago)
  Interventions: Other: Institutional standard of care; Other: Biosamples of airway and blood

INTERVENTIONS:
Other: Institutional standard of care — Institutional standard of care may involve the use of LungRADS (screening setting) or Fleischner criteria (either combined 2005, 2013 or 2017 guidelines)
Other: Biosamples of airway and blood — Identify biomarkers in biosamples from airway and blood for the preclinical detection of lung cancer.

SUMMARY:
DECAMP 1 PLUS aims to improve the efficiency of the diagnostic evaluation of patients with indeterminate pulmonary nodules (8-25 mm). Molecular biomarkers for lung cancer diagnosis measured in minimally invasive and non-invasive biospecimens may be able to distinguish between malignant or benign indeterminate pulmonary nodules in high-risk smokers. Ultimately, this study aims to validate molecular as well as clinical and imaging biomarkers of lung cancer in individuals with indeterminate lung nodules.

DETAILED DESCRIPTION:
The Detection of Early lung Cancer Among Military Personnel (DECAMP) consortium is a multidisciplinary and translational research program that previously initiated the DECAMP-1 and DECAMP-2 studies for lung cancer early detection. Now, with the support of Johnson and Johnson, 3 Veterans Administration Hospitals (VAH), 3 Military Treatment Facilities (MTF) and 12 academic hospitals as clinical study sites, several molecular biomarker laboratories, along with Biostatics, Bioinformatics, Pathology and Biorepository cores, we are expanding our work in lung cancer early detection.

ELIGIBILITY:
Inclusion Criteria:

* Radiologic diagnosis of solid indeterminate pulmonary nodule (0.8 to 2.5 cm) identified in the past 3 months OR semi-solid (mixed density) nodule with solid component of at least 0.6 cm identified in the past 12 months; must be of appropriate size at enrollment.
* CT scan completed within 3 months prior to enrollment
* Able to tolerate all biospecimen collection as required by protocol
* Able to comply with standard of care follow up visits including clinical exams, diagnostic work-ups, and imaging for approximately three years from enrollment
* Able to complete the Patient Lung History questionnaire with study staff

Arm 1 - Screening

* Age 55-77 years old
* Current and former smokers with 30 pack-years or more(and quit less than 15 years ago)

Arm 2 - Incidental

* Age > 45 years old
* Current and former smokers with 10 pack-years or more(and quit less than 15 years ago)

Exclusion Criteria:

* History or previous diagnosis of primary lung cancer, metastatic lung cancer, or any other non-lung cancer within 5 years (not including non-melanoma skin cancer)
* Symptoms of lung cancer (unexplained weight loss 10 lbs or more in 3 months, recent hemoptysis)
* Diagnosis of pure ground glass opacities for the target lesion on chest CT within the last 12 months (i.e., mixed features on the target lesion and pure ground glass opacity on non-target lesions are acceptable as mentioned above)

Min Age: 46 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are identified for inclusion in the study based on the observation of a lung nodule on screening or incidentally found by routine chest CT scans, between 0.8-2.5 cm diameter or observation of a mixed density nodule in which the solid portion is 0.6-2.5 cm diameter. These patients are managed according to institutional standard of care. This may involve the use of LungRADS (screening setting) or Fleischner criteria (either combined 2005, 2013 or 2017 guidelines)
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of lung cancer | 3 years
  The number of new cases of lung cancer that developed divided by the population at risk.

CONTACTS AND LOCATIONS:
Overall Officials: Ehab Billatos, MD, Principal Investigator — Boston University; Denise Aberle, MD, Principal Investigator — University of California, Los Angeles; George Washko, MD, Principal Investigator — Brigham and Women's Hospital
Locations (19):
- United States (19):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - University of California Los Angeles, Los Angeles, California
  - VA Greater LA Healthcare System, Los Angeles, California
  - Naval Medical Center San Diego, San Diego, California
  - University of Iowa, Iowa City, Iowa
  - Walter Reed Army Medical Center, Bethesda, Maryland
  - VA Boston Healthcare System, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Cleveland Clinic, Cleveland, Ohio
  - American College of Radiology [Administrative Site], Philadelphia, Pennsylvania
  - University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Brown University [Administrative Site], Providence, Rhode Island
  - VA Tennessee Valley Healthcare System, Nashville, Tennessee
  - MD Anderson Cancer Center [Administrative Site], Houston, Texas
  - Naval Medical Center Portsmouth, Portsmouth, Virginia
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Undecided